CLINICAL TRIAL: NCT05888831
Title: A Phase 1/2 Study of BMS-986449 Alone and in Combination With Nivolumab in Participants With Advanced Solid Tumors
Brief Title: A Study of BMS-986449 With and Without Nivolumab in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA120-1001; 2023-503484-42 (EudraCT Number); U1111-1287-3575 (Registry Identifier: WHO)
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors
Keywords: BMS-986449; Nivolumab; Cancer; Solid Tumors; Non-Small Cell Lung Cancer (NSCLC); Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation: BMS-986449 monotherapy (Experimental)
  Interventions: Drug: BMS-986449
- Dose Escalation: BMS-986449 + nivolumab (Experimental)
  Interventions: Drug: BMS-986449; Drug: Nivolumab
- Dose Escalation: BMS-986449 monotherapy pharmacodynamic (PD) cohorts (Experimental)
  Interventions: Drug: BMS-986449

INTERVENTIONS:
Drug: BMS-986449 — Specified dose on specified days
Drug: Nivolumab — Specified dose on specified days
  Other Names: OPDIVO®; BMS-936558
  Arms: Dose Escalation: BMS-986449 + nivolumab

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BMS-986449 alone and in combination with nivolumab in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have a histologically or cytologically confirmed, advanced, unresectable/metastatic, solid malignancy (measurable by Response Evaluation Criteria in Solid Tumors [RECIST] v1.1), and have received, be refractory to, ineligible for, or intolerant of existing therapy(ies) known to provide clinical benefit for the condition of the participant.

  * Part 1A may have a solid malignancy of any histology.
  * Part 1B is restricted to participants with Non-small cell lung cancer (NSCLC).
  * Part 1C is restricted to participants with Triple-negative breast cancer (TNBC).
* Tumor biopsy must be obtained for all participants (unless medically precluded).

Exclusion Criteria:

* History of Grade ≥ 3 toxicity related to prior T-cell agonist or checkpoint inhibitor therapy (eg, anti-cytotoxic T-lymphocyte-associated antigen 4 [CTLA-4], or anti-PD- 1/programmed death-ligand 1 [PD-L1] treatment, or any other antibody or drug specifically targeting T-cell co-stimulation or other immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures.
* Current or recent (within 3 months of study intervention administration) gastrointestinal disease or gastrointestinal surgery (eg, intestinal/gastric/colon resection) that could impact the absorption of study intervention.
* Any significant acute or chronic medical illness which would interfere with study intervention or follow-up in the opinion of the investigator.

Other protocol-defined criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose-Limiting Toxicities (DLTs) | Up to approximately 4 years
Number of participants with Adverse Events (AEs) | Up to approximately 4 years
Number of participants with Serious Adverse Events (SAEs) | Up to approximately 4 years
Number of participants with AEs leading to discontinuation | Up to approximately 4 years
Number of deaths | Up to approximately 4 years

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to approximately 4 years
Time of maximum observed concentration within a dosing interval (Tmax) | Up to approximately 4 years
Area under the concentration-time curve within a dosing interval (AUC[TAU]) | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (4):
  - Local Institution - 0021, Los Angeles, California
  - Local Institution - 0007, New Haven, Connecticut
  - Local Institution - 0010, Hackensack, New Jersey
  - Local Institution - 0022, Lake Success, New York
- Belgium (2):
  - Local Institution - 0016, Brussels, Bruxelles-Capitale, Région de
  - Local Institution - 0017, Ghent, Oost-Vlaanderen
- France (3):
  - Local Institution - 0002, Villejuif, Paris
  - Local Institution - 0004, Marseille, Provence-Alpes-Côte d'Azur Region
  - Local Institution - 0003, Bordeaux
- Italy (4):
  - Local Institution - 0023, Rozzano, Milano
  - Local Institution - 0024, Siena, Tuscany
  - Local Institution - 0026, Bergamo
  - Local Institution - 0025, Roma
- Netherlands (2):
  - Local Institution - 0030, Amsterdam, North Holland
  - Local Institution - 0018, Groningen
- Spain (5):
  - Local Institution - 0015, Málaga, Andalusia
  - Local Institution - 0013, Badalona, Barcelona [Barcelona]
  - Local Institution - 0012, Pamplona, Navarre
  - Local Institution - 0014, Madrid
  - Local Institution - 0011, Madrid

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05888831.html